CLINICAL TRIAL: NCT04769076
Title: A Prospective Phase II Clinical Trial of Paclitaxel (Albumin-bound) Combined With Cisplatin, PD-1 Inhibitors and IMRT in the Treatment of Locally Advanced Nasopharyngeal Carcinoma
Brief Title: The Paclitaxel (Albumin-bound) Combined With Cisplatin, PD-1 Inhibitors and IMRT in the Treatment of Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yang Yang, Professor of medicine, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-241-02
Record Dates: First submitted 2021-01-25; First posted 2021-02-24 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Taxes; Cisplatin; Immune Checkpoint Inhibitors; sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel(Album-bound) (Experimental): Subjects will receive neoadjuvant therapy with paclitaxel (albumin-bound) combined with cisplatin and PD-1 inhibitor (sintilimab) as well as radical concurrent radiotherapy and chemotherapy.
  Interventions: Combination Product: Paclitaxel（Albumin-bound）

INTERVENTIONS:
Combination Product: Paclitaxel（Albumin-bound） — Three courses of albumin-bound paclitaxel combined with cisplatin and PD-1 monoclonal antibody neoadjuvant treatment followed by cisplatin combined with IMRT (intensity modulated conformal radiotherapy) concurrent radiotherapy and chemotherapy
  Other Names: Cisplatin; PD-1 inhibitor (sintilimab); Radiotherapy

SUMMARY:
The purpose of this study in to observe the effectiveness and safety of paclitaxel (albumin-bound type) combined with cisplatin, PD-1 inhibitor and IMRT in the treatment of locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This trial is a prospective, open, single-arm phase II clinical trial. The trial will enroll 40 patients with nasopharyngeal cancer stage III-IVA (UICC 8th edition). Subjects will receive paclitaxel (albumin-bound) combined with cisplatin and PD-1 inhibitor (sintilimab) neoadjuvant therapy and radical concurrent chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed differentiated non-keratinizing carcinoma and undifferentiated non-keratinizing carcinoma
* The stage is Ⅲ-ⅣA (UICC 8th edition)
* Initial treatment patients without anti-tumor therapy
* No history of other malignant tumors
* Male or female, aged 18~70 years old
* Sufficient liver and kidney function: total bilirubin ≤ upper limit of normal (ULN); AST and ALT ≤ 2.5 times ULN; alkaline phosphatase ≤ 5 times ULN; creatinine clearance ≥ 80 mL/min
* Sufficient blood function: neutrophil count (ANC) ≥2×109/L, platelet count ≥100×109/L and hemoglobin ≥9 g/dL
* No serious heart, lung, liver, kidney and other important organ dysfunction
* Karnofsky score ≥70 points
* No autoimmune diseases
* Sign informed consent

Exclusion Criteria:

* Has performed anti-tumor treatment, including chemotherapy, radiotherapy, and surgery
* Discovery of distant metastases before treatment
* Receive live attenuated vaccine within 4 weeks before enrollment or plan to receive live attenuated vaccine during the study period
* Active, known or suspected autoimmune diseases
* Known history of primary immunodeficiency
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Women who are pregnant or breastfeeding
* Disagree to sign the informed consent form
* Patients who cannot cooperate with regular follow-up due to psychological, social, family and geographic reasons
* Simultaneously accept experimental treatment of other clinical research (in the treatment period of clinical research)
* Known allergic to possible chemotherapy drugs
* Accompanied by serious uncontrollable infections or medical diseases
* Major organ dysfunction, such as decompensated heart, lung, kidney, and liver failure, unable to tolerate radiotherapy and chemotherapy
* Laboratory examination: total bilirubin>upper limit of normal (ULN); AST and/or ALT>1.5 times ULN and accompanied by alkaline phosphatase>2.5 times ULN

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 month after the end of all treatments
  According to European Solid Tumor Efficacy Evaluation Standard (RECIST)